CLINICAL TRIAL: NCT00000198
Title: Piracetam for Treatment of Cocaine Addiction
Brief Title: Piracetam for Treatment of Cocaine Addiction - 3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kyle Kampman, Principal Investigator, University of Pennsylvania
Purpose: Treatment
Other Study IDs: NIDA-00238-3; K20DA000238 (NIH); K02-00238-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2013-12

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Piracetam

INTERVENTIONS:
Drug: Piracetam

SUMMARY:
The purpose of this study is to evaluate the effects of IV cocaine administration in cocaine dependent subjects maintained on piracetam while they are residing in an inpatient addictions treatment research unit and to subsequently follow these patients in an eight week open label assessment of piracetam in an outpatient treatment program.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-10; Primary Completion 1997-10 (Actual); Study Completion 1997-10 (Actual)

PRIMARY OUTCOMES:
Pulse, blood pressure
Adverse effects
High, anxiety, withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Kampman, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States